CLINICAL TRIAL: NCT03033498
Title: A Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of 24 Hour and 72 Hour Subcutaneous Infusions of ABBV-951 in Subjects With Parkinson's Disease
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Subcutaneous Infusions of ABBV-951 in Subjects With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M15-738
Record Dates: First submitted 2017-01-25; First posted 2017-01-26 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Parkinson's Disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- ABBV-951 Dose 1 (Experimental): Participants will receive dose 1 of ABBV-951.
  Interventions: Drug: ABBV-951
- ABBV-951 Dose 2 (Experimental): Participants will receive dose 2 of ABBV-951.
  Interventions: Drug: ABBV-951
- ABBV-951 Dose 3 (Experimental): Participants will receive dose 3 of ABBV-951.
  Interventions: Drug: ABBV-951
- ABBV-951 Dose 4 (Experimental): Participants will receive dose 4 of ABBV-951.
  Interventions: Drug: ABBV-951
- ABBV-951 Dose 5 (Experimental): Participants will receive dose 5 of ABBV-951.
  Interventions: Drug: ABBV-951
- ABBV-951 Dose 6 (Experimental): Participants will receive dose 6 of ABBV-951.
  Interventions: Drug: ABBV-951
- ABBV-951 Dose 7 (Experimental): Participants will receive dose 7 of ABBV-951.
  Interventions: Drug: ABBV-951
- ABBV-951 Dose 8 (Experimental): Participants will receive dose 8 of ABBV-951.
  Interventions: Drug: ABBV-951

INTERVENTIONS:
Drug: ABBV-951 — ABBV-951 administered by subcutaneous infusion.

SUMMARY:
The purpose of the study is to assess the safety, tolerability, and pharmacokinetics of single, ascending doses of ABBV-951 administered as a subcutaneous bolus infusion followed by a continuous subcutaneous infusion in subjects with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of definite idiopathic PD, which is LD responsive, according to the United Kingdom Parkinson's Disease Society Brain Bank Criteria.
* Subject must be taking an optimized and stable regimen of oral medications for PD, which has remained stable and unchanged for at least 30 days before dosing in this study. This regimen must include oral carbidopa/levodopa (CD/LD) tablets (e.g., Sinemet).
* Females must have negative results for pregnancy tests at screening and prior to confinement.
* If male, subject must be surgically sterile or practicing an adequate method of birth control from initial study drug administration until 30 days after last dose of study drug.
* Body Mass Index (BMI) is 18.0 to 38.0, inclusive.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* Receipt of any drug by injection within 30 days or within a period defined by 5 half-lives, whichever is longer, prior to study drug administration.
* History of significant skin conditions or disorders (e.g., psoriasis, atopic dermatitis, etc.) or evidence of recent sunburn, acne, scar tissue, tattoo, open wound, branding, or colorations that in the Investigator's opinion would interfere with the infusion of the study drug or could interfere with study assessments.
* Use of any medication from the prohibited concomitant therapies.
* Subjects with glomerular filtration rate (GFR) less than 45 ml/min/1.73 m2 as determined by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation.
* Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to initial study drug administration.
* Consideration by the investigator for any reason that the subject is an unsuitable candidate to receive ABBV-951.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-06-08 (Actual); Study Completion 2019-06-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Levodopa | Hour 0-24
  Maximum observed plasma concentration of levodopa following a single infusion of ABBV-951.
Time to maximum observed plasma concentration (Tmax) of Levodopa | Hour 0-24
  Time to maximum observed plasma concentration of levodopa following a single infusion of ABBV-951.
Area Under the Plasma Concentration-Time Curve (AUC) of Levodopa | Hour 0-24
  Area under the plasma concentration-time curve following a single infusion of ABBV-951.
Adverse Events | 24 hours
  Number of participants reporting adverse events
Terminal phase elimination rate constant (β) | Up to 72 hours
  Apparent terminal phase elimination rate constant (β or Beta)
Terminal phase elimination half-life (T1/2) | Up to 72 hours
  Terminal phase elimination half-life (t1/2) will be assessed.

SECONDARY OUTCOMES:
Corrected QT (QTc) Interval | Up to 76 hours
  QT interval adjusted for heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (7):
- United States (7):
  - Glendale Adventist Medical Ctr /ID# 166512, Glendale, California
  - Bioclinica Research - Orlando /ID# 169687, Orlando, Florida
  - Acpru /Id# 154976, Grayslake, Illinois
  - University of Kentucky Chandler Medical Center /ID# 169086, Lexington, Kentucky
  - Parexel Baltimore /ID# 169255, Baltimore, Maryland
  - QUEST Research Institute /ID# 166035, Farmington Hills, Michigan
  - Carolina Phase I, LLC /ID# 166034, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M15-738#additional-resources-section